CLINICAL TRIAL: NCT07134218
Title: A National Multicenter, Prospective, Randomized Controlled Study of Serplulimab Injection Combined With Bevacizumab to Improve the Complete Response Rate of Neoadjuvant Therapy for Locally Advanced Stage Intermediate and Low Rectal Cancer
Brief Title: Neoadjuvant Chemoradiotherapy Combined With Immunotherapy and Anti-angiogenesis in Treating Locally Advanced Rectal Cancer
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHOICE IV
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neoadjuvant chemoradiation therapy + serplulimab + bevacizumab (Experimental)
  Interventions: Drug: serplulimab、bevacizumab
- neoadjuvant chemoradiation therapy (Other)
  Interventions: Drug: serplulimab、bevacizumab; Other: neoadjuvant chemoradiation therapy

INTERVENTIONS:
Drug: serplulimab、bevacizumab — short-course radiotherapy 25 Gy in 5 fractions → 2-week break → 2 cycles of FOLFOX + serplulimab + bevacizumab → 2 cycles of FOLFOX + serplulimab.
Other: neoadjuvant chemoradiation therapy — short-course radiotherapy 25 Gy in 5 fractions → 2-week break → 4 cycles of FOLFOX alone.
  Arms: neoadjuvant chemoradiation therapy

SUMMARY:
This is a multicenter, prospective, randomized phase II trial designed to evaluate the efficacy and safety of short-course neoadjuvant chemoradiotherapy combined with the PD-1 monoclonal antibody serplulimab and the anti-angiogenic agent bevacizumab in patients with previously untreated pMMR/MSS middle and low locally advanced rectal cancer. The study plans to enroll a total of 200 participants (100 in the experimental arm and 100 in the control arm).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent to voluntarily participate in the study;
* Aged 18 to 75 years, inclusive, regardless of sex;
* Histologically confirmed rectal adenocarcinoma with immunohistochemistry results showing proficient mismatch repair (pMMR) or molecular testing results indicating microsatellite stability (MSS);
* Clinical baseline staging assessed by MRI as T3-4N0M0/TanyN+M, with negative mesorectal fascia (MRF);
* Tumor lower margin ≤7 cm from the anal verge;
* Surgically resectable;
* Capable of swallowing tablets normally;
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-1;
* No prior anti-tumor treatment for rectal cancer, including radiotherapy, chemotherapy, or surgery;
* Planned to undergo surgical treatment after completion of neoadjuvant therapy;
* No contraindications to surgery;
* Normal function of major organs.

Exclusion Criteria:

* History of allergy to any component of bevacizumab, serplulimab, 5-FU, or oxaliplatin.
* Prior or ongoing treatment with any of the following:

  1. Any tumor-targeted surgery, radiotherapy, chemotherapy, targeted therapy, or immunotherapy.
  2. Immunosuppressive drugs or systemic corticosteroid therapy for immunosuppressive purposes within 2 weeks before the first administration of the study drug (dose > 10 mg/day prednisone or equivalent). Inhaled or topical corticosteroids and adrenal corticosteroid replacement therapy (dose > 10 mg/day prednisone or equivalent) are permitted in the absence of active autoimmune disease.
  3. Live-attenuated vaccine within 4 weeks before the first administration of the study drug.
  4. Major surgery or severe trauma within 4 weeks before the first administration of the study drug.
* Presence of any active autoimmune disease or history of autoimmune disease, including but not limited to: interstitial pneumonia, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (participants on hormone replacement therapy may be considered for inclusion). Participants with psoriasis or childhood asthma/allergy that has fully resolved and requires no intervention in adulthood may be considered for inclusion, but those requiring bronchodilator therapy are not eligible.
* History of immunodeficiency, including HIV positivity, or other acquired or congenital immunodeficiency diseases, or history of organ transplant or allogeneic bone marrow transplant.
* Uncontrolled cardiac symptoms or diseases, including but not limited to: (1) NYHA class II or higher heart failure, (2) unstable angina, (3) myocardial infarction within the past year, (4) clinically significant supraventricular or ventricular arrhythmias that are not controlled or remain poorly controlled after clinical intervention.
* Severe infection (CTCAE > grade 2) within 4 weeks before the first administration of the study drug, such as severe pneumonia, bacteremia, or infection with complications requiring hospitalization. Baseline chest imaging showing active pulmonary inflammation, or presence of signs and symptoms of infection or need for oral or intravenous antibiotic therapy within 14 days before the first administration of the study drug (excluding prophylactic antibiotic use). History of active pulmonary tuberculosis infection identified through medical history or CT scan, or history of active pulmonary tuberculosis infection within the past year, or history of active pulmonary tuberculosis infection more than 1 year ago that was not properly treated.
* Active hepatitis B (HBV DNA ≥ 2000 IU/mL or 10⁴ copies/mL), hepatitis C (positive HCV antibody and HCV RNA above the lower limit of detection of the assay).
* Diagnosis of other malignancies within 5 years before the first administration of the study drug, unless the malignancy has a low risk of metastasis or death (5-year survival rate > 90%), such as adequately treated basal cell carcinoma or squamous cell carcinoma of the skin or cervical carcinoma in situ, which may be considered for inclusion.
* Pregnant or breastfeeding women.
* Presence of other factors that, in the investigator's judgment, may lead to forced discontinuation of the study, such as other severe diseases (including psychiatric conditions) requiring concomitant treatment, alcoholism, drug abuse, family or social factors that may affect the participant's safety or compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
The rate of cCR | 2 years
  Rate of patients who achieve clinical complete response

SECONDARY OUTCOMES:
Major Pathological Response | 2 years
  Rate of major pathological response assessed by postoperative pathology
Objective Response Rate | 2 years
  Objective response rate assessed by RECIST 1.1 criteria
Disease-Free Survival (DFS) | 2 years
  DFS was defined as the duration from the date of randomization to the date of the first recurrence (local, distant, or mixed) or death.
Overall Survival (OS) | 2 years
  Time from randomization to death due to any cause
Organ Preservation Rate (OPR) | 2 years
  Proportion of patients who achieve organ preservation by choosing a watch-and-wait strategy or local excision after attaining clinical or pathological complete response
Neoadjuvant Rectal Score (NAR) | 2 years
  Neoadjuvant rectal score assessed by postoperative pathology
Quality of Life Score (QoL) | 2 years
  Quality of life score during treatment and follow-up
Safety and Tolerability | 2 years
  Incidence of adverse events (AEs), incidence of abnormal laboratory values, and dose adjustments during treatment and follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Colorectal Surgery in Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD would be available upon reasonable request.
Supporting Information: Study Protocol
Time Frame: 2 years